CLINICAL TRIAL: NCT04343404
Title: STUDY ECMO-COVID-19 : Place of ECMO in the Management of Severe Refractory ARDS Associated With Covid-19
Brief Title: Place of ECMO in the Management of Severe Refractory ARDS Associated With Covid-19
Acronym: ECMO-COVID-19
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7772
Record Dates: First submitted 2020-04-08; First posted 2020-04-13 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2020-04

CONDITIONS: Respiratory Distress Syndrome
Keywords: Respiratory Distress Syndrome; ARDS; SARS-COV-2; Extracorporeal membrane oxygenation; ECMO; Veno-venous ECMO
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Describe COVID-19 patients who are receiving ECMO-VV respiratory replacement and what happens to them.

ELIGIBILITY:
Inclusion Criteria:

* Patient over the age of 18;
* Diagnostic COVID-19 by RT-PCR;
* Hospitalisation in resuscitation for the management of complications related to COVID-19
* Implanted ECMO-VV during hospitalisation;
* Patient agreeing to participate in the study

Exclusion Criteria:

* Sujet under guardianship or trusteeship
* Sujet under safeguard of justice

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients with a COVID-19 diagnosis by RT-PCR
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-04-15 (Actual)

PRIMARY OUTCOMES:
Retrospective description of COVID-19 patients receiving respiratory ECMO-VV supplementation and what happens to them | Files analysed retrospectily from March 1st, 2020 to April 15, 2020 will be examined

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Emmanuel FALCOZ, MD, PhD, Study Director — Service de Chirurgie Thoracique Nouvel Hôpital Civl Hôpitaux Univesitaires de Strasbourg
Locations (1):
- Service de Chirurgie Thoracique Nouvel Hôpital Civil Hôpitaux Universitaires de Strasbourg, Strasbourg, France